CLINICAL TRIAL: NCT01873651
Title: The Reverse Delta III Total Shoulder Prosthesis - Longerm Results in 98 Patients
Brief Title: Longterm Outcome of the Delta III Inverse Prosthesis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study has been withdrawn due to too few patients
Sponsor: Schulthess Klinik (Other)
Responsible Party: Principal Investigator, Matthias Flury, Principal Investigator (Department of Upper Extremity), Schulthess Klinik
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Delta III
Record Dates: First submitted 2013-06-05; First posted 2013-06-10 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Rotator Cuff Tear Arthropathy
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Delta III (Experimental): Implantation of a Delta III Prosthesis
  Interventions: Device: Implantation of a Delta III Prosthesis

INTERVENTIONS:
Device: Implantation of a Delta III Prosthesis — Implantation of a Delta III Prosthesis

SUMMARY:
The aim of the study is to describe the results after > 10 years due to a prosthesis implant.

DETAILED DESCRIPTION:
The aim of the study is to measure the gain of the benefit in function an painreduction which the patient yields with this type of prosthesis in a longterm (> 10 years )outcome. Additionally the long-term results will be compared with the mid-term results and the literature. Furthermore the complications since the mid-term measurement time point will be determined.

ELIGIBILITY:
Inclusion Criteria:

* implantation of a Delta III - prothesis
* timeframe (Oct 1998 - Dec 2002)
* delta-pectoral approach
* written informed consent

Exclusion Criteria:

* Implantation because of a revision
* Complaints, which make it difficult to follow instructions or even prevent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Constant Murley Score | 10 years

SECONDARY OUTCOMES:
cASES | 10 years
pASES | 10 years
SF-36 | 10 years
DASH-Questionannaire | 10 years
SPADI | 10 years
x-ray (Sperling Classification) | 10 years
x-ray (Sirveaux Classification) | 10 years
Description of the glenoid | 10 years
  Description of the situation:
  e.g.
  * any dissociation of the gleonid
  * any migration of the glenoid
Description of the stem | 10 years
  Description of the situation:
  e.g.
  - change of the position

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Flury, Dr., Principal Investigator — Schulthess Klinik, Upper Extremities Department